CLINICAL TRIAL: NCT06422689
Title: ANCHOR - Assessment of Combination Short-Acting BroNchodilator and Inhaled Corticosteroid Rescue Therapy on Health Outcomes in Routine Care
Brief Title: Combination Short-Acting BroNchodilator and Inhaled Corticosteroid Rescue Therapy on Health Outcomes in Routine Care
Acronym: ANCHOR
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Premier HealthCare Solutions Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6930L00001
Record Dates: First submitted 2024-04-10; First posted 2024-05-21 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Effectiveness; Asthma; Exacerbation; Healthcare resource utilization; Cost; Albuterol/budesonide; Short-acting beta-agonist (SABA); Inhaled corticosteroids (ICS); Rescue; Switch; Oral corticosteroid; Patients reported asthma symptoms; PT027
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Albuterol and budesonide inhalation aerosol (Experimental): Participants will receive a fixed-dose combination of albuterol (90mcg) and budesonide (80mcg) administered as 2 inhalations (180mcg/160mcg) via pressurized metered dose inhaler (pMDI) as needed for asthma symptoms, for up to 12 inhalations (6 doses) in a 24-hour period.
  Interventions: Drug: Albuterol and budesonide inhalation aerosol

INTERVENTIONS:
Drug: Albuterol and budesonide inhalation aerosol — Participants will receive a fixed-dose combination of albuterol (90mcg) and budesonide (80mcg) administered as 2 inhalations (180mcg/160mcg) via pressurized metered dose inhaler (pMDI) as needed for asthma symptoms, for up to 12 inhalations (6 doses) in a 24-hour period.
  Other Names: PT027

SUMMARY:
ANCHOR is a prospective, phase IV, interventional, single-arm, open-label study of 1,500 adult participants with symptomatic asthma requiring the use of rescue therapy aimed to compare the asthma exacerbation rates before and after switching from albuterol or levalbuterol to albuterol plus budesonide inhalation aerosol as rescue therapy.

DETAILED DESCRIPTION:
This study will primarily compare rates of asthma exacerbation during 12-month pre-switch period and 12-month post switch period among participants with asthma needing a rescue therapy. Other outcomes of interest for comparison between the pre- and post-switch periods include asthma-related oral corticosteroids (OCS) use, asthma exacerbation-related hospitalizations, emergency department (ED) visits, urgent care visits, outpatient visits, telehealth visits, and asthma-related and asthma exacerbation-related healthcare costs. The use of asthma control and rescue medications will be collected to understand treatment patterns in the real-world US context.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above as of enrollment date.
2. At least 1 diagnosis of asthma prior to the enrollment date documented in patient record.
3. At least 1 prescription filled for Short-acting beta-agonist (SABA)-only inhaler (i.e., albuterol-only or levalbuterol only inhalers) within 12 months before enrollment date.
4. At least 1 severe asthma exacerbation within 12 months before enrollment date.
5. Had both medical and pharmacy insurance coverage (e.g., Medicare, Medicaid, and commercial insurance) for at least 12 months before enrollment date and without foreseeable plans to discontinue insurance coverage within 12 months after enrollment date.
6. Participants also need to meet each of the following inclusion criteria:

   1. Willingness to use albuterol and budesonide as rescue as instructed by their physician, prescribing information, and United States instruction for use (USIFU).
   2. Willingness to respond to quarterly safety inquiries.
   3. Willingness to participate in quarterly electronic patient-reported outcome (PRO) surveys via email or text.
   4. Physician decision that participant is eligible for treatment with albuterol and budesonide as rescue according to the approved United States prescribing information (USPI).

Exclusion Criteria:

1. Conditions with major respiratory diagnoses including chronic obstructive pulmonary disease (COPD), cystic fibrosis, pulmonary fibrosis, bronchiectasis, respiratory tract cancer, bronchopulmonary dysplasia, sarcoidosis, lung cancer, interstitial lung disease, pulmonary hypertension, and tuberculosis in 12 months before the enrollment date.
2. Inpatient admission or emergency department or urgent care visit due to asthma in the 10 days before enrollment date, or self-reported use of systemic corticosteroid for the treatment of asthma in the 10 days before enrollment date. Participants who were screen-failed due to this criterion may be re-screened once the participant is more than 10 days post asthma-related inpatient admission, emergency department or urgent care visit, or systemic corticosteroid use.
3. Chronic use of oral corticosteroids (for any condition) within 3 months before enrollment date. Chronic use of oral corticosteroids is defined as: daily or every other day use for 21 days or longer.
4. History of albuterol and budesonide as rescue use within 12 months before enrollment date.
5. History of any malignancy (except non-melanoma neoplasms of skin) in 12 months before the enrollment date.
6. For females only - currently pregnant or breastfeeding on enrollment date. Participants are excluded from the study if any of the following criteria apply.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1507 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2026-04-29 (Estimated)

PRIMARY OUTCOMES:
Asthma exacerbation | During 12-month pre-switch and 12-month post-switch periods
  Annualized Severe Asthma exacerbation rate

SECONDARY OUTCOMES:
Asthma exacerbation-related HCRU | During 12-month pre-switch and 12-mont post switch periods
  Percentage of patients with Asthma exacerbation-related HCRU
Asthma exacerbation-related cost | During 12-month pre-switch and 12-month post-switch periods
  Asthma exacerbation-related cost in US Dollars
Asthma-related cost | During 12-month pre-switch and 12-month post-switch periods
  Asthma-related cost in US Dollars
Asthma- related Oral Corticosteroid (OCS) use | During 12-month pre-switch and 12-month post-switch periods
  Mean number of Asthma- related Oral Corticosteroid (OCS) prescriptions
Change in asthma exacerbation-related HCRU at health system level | During 12-month pre-switch and 12-month post-switch periods
  Percentage of patients with Asthma exacerbation-related HCRU at the health system level

OTHER OUTCOMES:
Improvement in patient reported asthma symptoms and treatment satisfaction using the ANCHOR PRO Questionnaire | at 3-, 6-, 9-, and 12-month post-switch
  Percentage of patients who reported improvement in asthma symptoms and satisfaction with albuterol and budesonide treatment as rescue therapy
Asthma-related controller and rescue medication use | During 12-month pre-switch and 12-month post switch periods separately
  Number of fills of asthma-related controllers and rescue medications
Experience of (yes/no) and number of safety events | During 12-month post-switch period
  Number of adverse events (AE) and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Research Site, North Hollywood, California
  - Research Site, Walnut Creek, California
  - Research Site, Louisville, Kentucky
  - Research Site, Boston, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Asheville, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, DuBois, Pennsylvania
  - Research Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/